CLINICAL TRIAL: NCT03221140
Title: Observational Study About the Feasibility, Safety and Efficacy of Outpatient Parenteral Antimicrobial Therapy (OPAT)
Brief Title: Outpatient Parenteral Antimicrobial Therapy (OPAT)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Serge de Valliere, MD,MSc, Principal Investigator, University of Lausanne Hospitals
Other Study IDs: 34/14
Record Dates: First submitted 2017-06-27; First posted 2017-07-18 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Outpatient parenteral antimicrobial therapy — Administration of intravenous antimicrobials on an outpatient basis
  Other Names: OPAT

SUMMARY:
Outpatient parenteral antimicrobial therapy (OPAT) has been recognised as a useful, cost-effective and safe alternative to inpatient treatment, but no formal OPAT unit existed in Switzerland until recently. In December 2013 an OPAT unit was established at Lausanne University Hospital. The investigators plan to investigate the efficacy, safety and economicity of outpatient parenteral antimicrobial therapy administered at the new OPAT unit of the Lausanne University Hospital starting in January 2014 until December 2020.

DETAILED DESCRIPTION:
Some patients require parenteral antibiotic therapy, but are well enough to return home. Outpatient parenteral antimicrobial therapy (OPAT) was first developed in the USA in the 1970s for patients with cystic fibrosis, before being adopted by other countries. It has been recognised as a useful, cost-effective and safe alternative to inpatient treatment. It is now a standard care in several countries and different national guidelines have been established. There are various models of care for OPAT and most OPAT centres provide hospital-centred nursing programmes or services based on nurses visiting the patient's home. A few centres have also shown that self-administration of intravenous antibiotic therapy is an effective and safe option for selected patients. Furthermore, use of continuous infusion of antibiotics increases the number of feasible treatments. Continuous infusion by pumps of antibiotics with a time-dependent killing mechanism is a practical option which has been described. In Europe, even if many infectious disease specialists feel that OPAT is required, it is still underdeveloped because of lack of funding, lack of leadership and lack of coordination between hospitals and community care.

In the last decades, programs to enhance care delivery on an outpatient basis in order to contain health costs have been developed in Switzerland. However administration of outpatient intravenous antibiotic therapy for patients who require parenteral therapy, but are otherwise fit enough to go home, hasn't been used widely until recently. In December 2013, an outpatient parenteral antibiotic treatment (OPAT) unit was initiated at Lausanne University Hospital with the goal of offering an alternative treatment programme that is equally effective and as safe as inpatient treatment.

The purpose of this study will be to investigate the efficacy, safety and economicity of treatments administered at the new OPAT unit of the University Hospital of Lausanne in the context of the Swiss Health System.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the OPAT unit of Lausanne University Hospital

Exclusion Criteria:

* Unable to give informed consent
* Refusing participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to the OPAT unit of Lausanne Unversity Hospital
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2014-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of treatment outcomes | 2014-2020
  Efficacy of OPAT will be evaluated by recording the treatment outcome. Patients will be categorized 3 months after end of treatment as cured, as treatment failure or as a relapse according to the following definitions:
  * cured: absence of fever and no clinical sign of the site of infection.
  * treatment failure: patient readmitted to hospital because of infection related complications
  * relapse: patients considered as cured at the end of OPAT, but who had again signs of infection at the same site within 3 months after end of OPAT.
Evaluation of the incidence of adverse events | 2014-2020
  Evaluation of the safety of OPAT will be done by measuring the rate of adverse events and their severity during OPAT. All adverse events will be recorded and classified according to their severity according the grade classification (grade 1 to 5) as recommended by the Common Terminology Criteria for Adverse Events (CTCAE). (https://evs.nci.nih.gov/ftp1/CTCAE/CTCAE_4.03_2010-06-14_QuickReference_5x7.pdf)
Economic evaluation | 2014-2020
  The cost of outpatient parenteral antimicrobial treatments will be estimated and compared to similar economic evaluations of other centres published in the literature.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Outpatient Care and Community Medicine, University Hospital of Lausanne, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Voumard R, Gardiol C, Andre P, Arensdorff L, Cochet C, Boillat-Blanco N, Decosterd L, Buclin T, de Valliere S. Efficacy and safety of continuous infusions with elastomeric pumps for outpatient parenteral antimicrobial therapy (OPAT): an observational study. J Antimicrob Chemother. 2018 Sep 1;73(9):2540-2545. doi: 10.1093/jac/dky224. PMID 29982449